CLINICAL TRIAL: NCT07277387
Title: A Multicenter Prospective Observational Study on the Plasma Proteomic Profiling of Human and Microbial Proteins for the Early Identification of Biomarker Combinations (Combitypes) Associated With Complications in Oncohematologic Patients With Febrile Neutropenia
Brief Title: Plasma Host-Microbe Proteomics to Predict Complications in High-risk Febrile Neutropenia
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Other Study IDs: COMBITYPES-FN
Record Dates: First submitted 2025-11-18; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-10

CONDITIONS: Febrile Neutropenia
Keywords: febrile neutropenia; hematologic malignancy; proteomics; sepsis; biomarkers; septic shock; mass spectrometry
MeSH Terms: conditions — Febrile Neutropenia; Hematologic Neoplasms; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Whole blood (10 mL) will be collected in EDTA tubes at two time points: (1) at fever onset before the initiation of empirical antibiotic therapy and (2) 48 hours later. Plasma will be separated by centrifugation, aliquoted, and stored at -80°C until proteomic analysis.
  In addition to plasma, residual buffy coat fractions will be retained for DNA extraction to enable future genomic or metagenomic studies related to host or microbial signatures.
  All biospecimens will be pseudonymized and stored at the BioSepsis Laboratory (IBSAL) and subsequently transferred to the CAUSA Biobank for long-term storage and controlled access.
  Samples will be registered in the Spanish National Biobank Registry, and their use in future studies will require approval by the relevant Research Ethics Committee.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-risk FN cohort: Adult onco-hematologic inpatients meeting inclusion criteria; two plasma draws at fever onset and 48 h.
  Interventions: Biological: Plasma and DNA sample collection for proteomic and genomic analysis

INTERVENTIONS:
Biological: Plasma and DNA sample collection for proteomic and genomic analysis — Collection of 10 mL of peripheral blood in EDTA tubes at fever onset (before antibiotic initiation) and 48 hours later for proteomic and genomic analysis. Samples are processed to obtain plasma and DNA, which will be used for mass spectrometry-based proteomics and potential metagenomic studies.

SUMMARY:
Febrile neutropenia (FN) is a common oncologic emergency in patients with hematologic malignancies, associated with high morbidity and mortality. Early identification of patients at higher risk of complications such as sepsis or septic shock is critical to optimize antimicrobial management.

This study aims to characterize the human and microbial plasma proteome using high-resolution mass spectrometry to identify biomarker combinations ("combitypes") capable of predicting complications in oncohematologic patients with FN.

A cohort of 350 adult patients with high-risk FN and initially uncomplicated clinical presentation will be enrolled across three tertiary hospitals. Plasma samples will be collected at fever onset (before antibiotic initiation) and after 48 hours. Proteomic data will be integrated with clinical information using multivariate and machine learning models to develop a predictive model for complications.

DETAILED DESCRIPTION:
This multicenter, prospective, observational study will evaluate whether combined proteomic profiles of host and microbial origin can predict complications in patients with hematologic malignancies presenting with high-risk febrile neutropenia (FN).

FN is defined as an oral temperature ≥38.3 °C once or ≥38.0 °C for ≥1 hour in patients with an absolute neutrophil count (ANC) <500 cells/mm³ or expected to decrease below that threshold within 48 hours. Despite empirical broad-spectrum antibiotics, up to 50% of these patients develop sepsis, and 10% progress to septic shock.

Current biomarkers such as C-reactive protein (CRP) or procalcitonin (PCT) have limited specificity in this immunocompromised population. This study proposes a novel integrative proteomic approach based on mass spectrometry to simultaneously quantify host and microbial proteins in plasma, identifying molecular patterns associated with poor outcomes.

Plasma samples (10 mL, EDTA) will be obtained at two time points: the first febrile episode (prior to antibiotic administration) and 48 hours later. Proteins will be processed using PreOmics® ENRICHplus technology and analyzed via LC-MS/MS on an Evosep One-timsTOF Pro2 platform. Differentially expressed proteins will be identified using a data-independent acquisition (DIA-PASEF) workflow and validated in a subset of 200 patients through targeted mass spectrometry.

Clinical, analytical, and microbiological data will be collected via the REDCap platform. Machine learning models (XGBoost, SHAP interpretability) will be used to generate a predictive risk model for complications, integrating proteomic and clinical data.

This study is expected to establish a new decision-support tool for early identification of high-risk FN patients, facilitating personalized antimicrobial strategies and improved prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Written informed consent provided by patient or legal representative.
* Diagnosis of hematologic malignancy under induction chemotherapy, post-allogeneic hematopoietic stem cell transplantation, or CAR-T therapy.
* High-risk febrile neutropenia (ANC ≤ 100 cells/mm³, expected duration ≥ 7 days, or significant comorbidities).
* Fever defined as oral temperature ≥38.3 °C once or ≥38.0 °C for ≥1 hour.
* Hospitalized or requiring immediate admission at the time of FN diagnosis.

  ´- Initial uncomplicated clinical presentation, with no previous infection or colonization by multidrug-resistant bacteria.
* Eligible for initial monotherapy with broad-spectrum empirical antibiotic.
* Availability for serial plasma sampling and clinical follow-up.

Exclusion Criteria:

* Age <18 years.
* Low-risk FN according to MASCC/CISNE criteria.
* Initial sample collected after antibiotic administration.
* Decline or inability to provide informed consent.
* Any condition preventing safe participation or reliable sample collection.
* Fever induced by noninfectious causes (considered as adjustment factor, not exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncohematologic Patients With Febrile Neutropenia
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Identification of plasma host-microbial proteomic signatures (combitypes) associated with major complications in febrile neutropenia. | Within 7 days from fever onset.
  Evaluation of proteomic profiles (human and microbial) associated with hemodynamic instability, sepsis, septic shock, or death.

SECONDARY OUTCOMES:
Dynamic changes in plasma proteome over 48 hours | 0-48 hours
  Assessment of longitudinal variations in host and microbial protein levels between baseline and 48 hours.
Predictive performance of identified combitypes versus conventional biomarkers (CRP, PCT) | Up to 7 days.
  Comparison of ROC-AUC for new proteomic models against current inflammatory markers.
Correlation between microbial proteomic profiles and microbiologically documented infections | During hospitalization (up to 30 days).
  Association between detected microbial peptides and confirmed pathogens.
Development of a predictive model for complications | Study duration (36 months).
  A predictive risk model for complications will be developed using machine-learning algorithms (XGBoost) based on the integration of plasma proteomic data and relevant clinical parameters collected at fever onset and during follow-up. The model will be trained and internally validated within the full study cohort using cross-validation techniques to optimize predictive performance and minimize overfitting.
Validation of selected protein biomarkers by targeted mass spectrometry | By end of study (month 36).
  Selected protein biomarkers previously identified through discovery-phase proteomic profiling will be validated using targeted LC-MS/MS mass spectrometry in plasma samples from 200 patients within the study cohort. This validation phase will assess the analytical performance (including reproducibility, accuracy, and sensitivity) of the selected biomarkers, as well as their clinical relevance in predicting complications such as hemodynamic instability, sepsis, septic shock, or death. This outcome cannot be divided into sepparate ones, as biomarker expression will be analyzed as a whole, given the fact that until the trial begins, the biomarkers associated with complications in oncohematologic patients with febrile neutropenia will be unkown. This outcome will determine the feasibility of implementing the identified biomarkers as prognostic tools in routine clinical practice for the early risk stratification of patients

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Francisco Bermejo Martín, MD PhD, Principal Investigator — Centro Asistencial Universitario de Salamanca (CAUSA)
Locations (3):
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Complejo Asistencial Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: Yes
Following anonymization, individual participant-level data supporting the publications will be made available. These data include demographic and clinical variables collected in REDCap. A data dictionary, eCRF, and-when possible-analysis scripts (R/Python) and FAIR-compliant metadata will also be provided.
  Data will be hosted within the controlled infrastructure of the project (XNAT/Core-lab) and, for controlled dissemination, within the Zenodo community of IBSAL, with DOI assignment and regulated access, in accordance with the GDPR/LOPDGDD and the study protocol as approved by the Research Ethics Committee.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available starting 12 months after publication of the primary results and will remain accessible for at least 5 years thereafter.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access. Requests will be reviewed by the study's Data Committee/Steering Committee. Applications should be addressed to the Principal Investigator (Jesús Francisco Bermejo Martín). A Data Use Agreement (DUA) will be required, including commitments to non-reidentification, appropriate data security, and mandatory citation of both the source and dataset DOI. Applicants may also be required to share their analytical code and a publication plan prior to authorization.